CLINICAL TRIAL: NCT07145580
Title: Clinical Application of a Combined Lactulose H2-breath Test With Abdominal Imaging to Assess the Digestive Function: a Retrospective Cohort Study
Brief Title: Combined Lactulose H2-breath Test With Abdominal Imaging
Status: Recruiting | Type: Observational
Sponsor: Klinik Arlesheim (Other)
Collaborators: Kantonsspital Baselland Bruderholz (Other)
Responsible Party: Sponsor
Other Study IDs: KlinikArlesheim
Record Dates: First submitted 2025-07-11; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Food Intolerance Syndromes; Small Intestinal Bacterial Overgrowth Syndrome (SIBO); Breath Tests
Keywords: Irritable bowel syndrome (IBS); Functional bloating; Functional Diarrhea; Food Intolerance Syndromes; Small intestinal bacterial overgrowth syndrome (SIBO); Hydrogen Breath Test
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for hydrogen breath testing: Adult patients referred for hydrogen breath testing between 2020 and 2024 were included in this cohort. All patients included in the analysis signed general consent for the use of anonymized clinical data in studies. Indications for investigation included assessment of causes of digestive symptoms or maldigestion. Patients had laboratory and other imaging or endoscopic investigations that showed no evidence of organic pathology.
  This retrospective cohort study reports the performance of a combined 20g lactulose H2 breath test with radiographic abdominal imaging to assess OCTT, SIBO, and carbohydrate tolerance. The novel innovation in this method is to confirm OCTT by taking an X-ray of the abdomen when H2 production increases during the examination. If contrast agent is NOT visible in the caecum when H2 increases, then SIBO is present. Otherwise, if contrast agent is present in the caecum, then results confirm OCTT and carbohydrate intolerance.

SUMMARY:
Hydrogen (H₂) breath tests serve several purposes. (i) detect malabsorption of carbohydrates such as lactose and fructose, (ii) measurement of oro-caecal transit time (iii) associate hydrogen production with the onset of abdominal symptoms like bloating, flatulence, pain, and diarrhea (which indicates carbohydrate intolerance), and (iv) diagnose small intestinal bacterial overgrowth (SIBO).

It is important to distinguish between carbohydrate intolerance and SIBO because their treatments differ significantly. Carbohydrate intolerance is typically managed through dietary restrictions, while SIBO requires antibiotic therapy. However, recent guidelines have questioned the accuracy of hydrogen breath tests in diagnosing SIBO due to variability in OCTT measurements. This limitation can be addressed by combining H₂ breath tests with imaging techniques such as scintigraphy, which independently confirm OCTT. When this combined approach is used, SIBO is diagnosed if the rise in breath H₂ occurs before the contrast agent appears in the large bowel. Despite its benefits, this combined method faces organizational and financial challenges that limit its routine clinical use.

This retrospective cohort study aims to assess the clinical performance of a cheap and simple test that combines a 20g lactulose H₂ breath test with simple radiographic abdominal imaging to assess OCTT, SIBO, and carbohydrate tolerance. The novel innovation in this method is to confirm oro-caecal transit by taking an X-ray of the abdomen when H₂ production increases during the examination. If the contrast agent is not visible in the cecum when H₂ rises, this indicates the presence of SIBO. Conversely, if the contrast agent is present in the cecum at that time, it confirms normal OCTT, and any abdominal symptoms occurring after this point support a diagnosis of carbohydrate intolerance.

If the method is proven to be valid, then this simple test will greatly facilitate the accurate diagnosis of SIBO and carbohydrate intolerance, allowing for more appropriate treatment decisions.

DETAILED DESCRIPTION:
Carbohydrate malabsorption can be detected by hydrogen (H2) breath tests because this gas is not generated by human cells but is derived exclusively through anaerobic fermentation of carbohydrates by enteric microflora. Increased concentrations of this biomarker in breath after oral ingestion of a fermentable carbohydrate indicates that this substrate has not been fully absorbed by the small bowel and has come into contact with saccharolytic bacteria.

Several substrates have been used in H2 breath tests. The aims of these tests include (I) detection of carbohydrate malabsorption of lactose and fructose and other substrates that are variably absorbed in the small bowel, (II) measurement of the time interval between ingestion of an unabsorbable carbohydrate, such as lactulose, and its contact with colonic bacteria in the cecum (oro-cecal transit time, OCTT), and (III) association of H2 gas production with onset of abdominal symptoms like bloating, flatulence, abdominal pain and diarrhea, i.e. carbohydrate intolerance (IV) diagnosis of small intestinal bacterial overgrowth (SIBO) by an "early rise" (e.g.; <90 minutes) in H2 after ingestion of a test substance (e.g. glucose or lactulose), due to abnormally high concentrations of bacteria in the small intestine.

The distinction between carbohydrate intolerance and SIBO is important because treatment of the two conditions is different. The former is most often managed by dietary restriction, whereas the latter is treated by antibiotics. Recent guidelines and editorials have questioned the accuracy of H2 breath tests in the detection of SIBO primarily due to high variation in measurements of OCTT. In particular, rapid OCTT leading to an early rise in H2 after ingestion of a substrate can lead to a false positive diagnosis of SIBO and treatment with inappropriate medication. This limitation can be addressed by combining H2 breath tests with scintigraphic imaging that provides an independent assessment of OCTT. When this methodology is applied, SIBO is diagnosed when there is an increase in breath H2 before scintigraphic contrast appears in the large bowel. However, there are important organizational and financial barriers to implementation of this approach in routine clinical practice.

This retrospective cohort study reports the performance of a cheap and simple test that combines a 20g lactulose H2 breath test with radiographic abdominal imaging to assess OCTT, SIBO, and carbohydrate tolerance. The novel innovation in this method is to confirm oro-caecal transit by taking an X-ray of the abdomen when H2 production increases during the examination. If contrast agent is NOT visible in the caecum when H2 increases, then SIBO is present. Otherwise, if contrast agent is present in the caecum, then results confirm OCTT and the occurrence of abdominal symptoms after this time is consistent with the diagnosis of carbohydrate intolerance.

The rationale of using 20g lactulose in this investigation is based on the results of a series of studies from the principle investigator and others that showed (i) H2 breath test results after ingestion of 20g lactulose are statistically not different to those after ingestion of 20g lactose in a patient with lactase deficiency. (ii) The 20g lactulose nutrient challenge test can identify patients with carbohydrate intolerance (i.e. lactulose is a representative FODMAP) especially in patients with visceral hypersensitivity, a common feature of patients with irritable bowel syndrome (IBS). (iii) a dose response relationship between the amount of substrate ingested and the likelihood of symptoms occurring in health and disease, with IBS patients statistically significantly more likely to have symptoms after ingestion of 20g indigestible carbohydrate compared to healthy controls (OR >3). (iv) pilot data that suggests patients with SIBO identified using combined 20g lactulose H2 breath test with abdominal imaging have more severe symptoms than patients with food intolerance without SIBO and also report an improvement in abdominal symptoms after treatment with a non-absorbable antibiotic (rifaximin) which does not occur in patients without SIBO.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for breath testing to assess the causes of digestive symptoms or maldigestion 2020-2024
* Patients signed general consent to allow use of clinical data obtained during clinical assessment and breath testing to be used in research project.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for breath testing to assess the causes of digestive symptoms or maldigestion 2020-2024
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Practicability and safety of the novel. concurrent 20g lactulose H2 breath test with abdominal imaging | 3 hours
  This pilot feasibility study will report the practicability and safety of the concurrent 20g lactulose H2 breath test with abdominal imaging, defined as:
  * Practicability / Technical success in performance of the investigation defined by (i) correct documentation of H2 production and patient symptoms using validated questionnaires (ii) timely acquisition of abdominal imaging within 20 min of H2 increase after test substance ingestion (both expressed as percentage ot total) .
  * Safety of the concurrent 20g lactulose H2 breath test with abdominal imaging, defined as the ability of patients (i) to ingest the test substrate (400ml) without nausea and vomiting (ii) to complete the 3-hour operating procedure without severe abdominal symptoms that require medical treatment and / or termination of test (both expressed as percentage ot total).
  The primary outcome measures are descriptive and not chosen to demonstrate superiority of this methodology compared to existing techniques.

SECONDARY OUTCOMES:
Inter-rater agreement of the oro-caecal transit time | 3-hours
  Assessment of oro-caecal transit time by radiography during 3-hour breath test study by clinician responsible for breath test procedure and also by radiologist reporting result of abdominal X-ray.
  Time is measured in minutes from ingestion of test substance. All cases assessed independently by two observers (gastroenterology, radiology).
  Agreement assessed by simple percent agreement and Cohen's kappa. Additionally, Cases in which there is disagreement as to whether contrast agent has arrived in the caecum will be reviewed by clinician, radiologist and principle investigator.
Assess prevalence of food intolerance and SIBO in patients referred for breath testing | 3-hours
  Describe the results obtained by the concurrent 20g lactulose H2 breath test with abdominal imaging in terms of the prevalence of SIBO and food intolerance in patients referred for breath testing. A planned sub-analysis of results in patients with clinical diagnosis of IBS compared to patients with other diagnoses will also be performed.

OTHER OUTCOMES:
Exploratory analysis of causes of abdominal symptoms during lactulose hydrogen breath test | 3-hours
  Correlation of demographic (age, sex) and clinical factors (specifically presence / absence of irritable bowel syndrome based on Rome IV classification), and physiological measurements of oro-caecal transit time (minutes) and Hydrogen gas production (ppm) with the occurrence of abdominal symptoms (assessed by validated 5 point Likert scale) will be assessed by Univariate and step-wise multivariate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Arlesheim, Arlesheim, Basel-Landschaft, Switzerland